CLINICAL TRIAL: NCT03303430
Title: Correlation Between Cerebral Microembolisation and Plaque Characteristics After Carotid Revascularization
Brief Title: Microembolisation After Carotid Revascularisation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Loraine Fisch, Principal investigator, University Hospital, Geneva
Other Study IDs: PLASTIS
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Carotid Stenosis
Keywords: cerebral microembolisation; plaque characteristics
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Surgery group: This patient's group will benefit from a endarteriectomy in order to treat their carotid stenosis.
  Interventions: Diagnostic Test: MRI
- Stenting group: This patient's group will benefit from a stenting of their carotid in order to treat their stenosis.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Diffusion weighted imaging 24 hours after revascularisation

SUMMARY:
Microembolisation identified on diffusion-weighted magnetic resonance imaging (DW-MRI) is recognized as an important outcome measure for carotid revascularization procedures such as carotid stenting (CAS) or carotid endarterectomy (CEA). In fact, cerebral microembolisation occurring during revascularization procedures is associated with an increased risk of peri- and post-procedural stroke, transient ischemic attack as well as neurocognitive decline. Carotid artery stenting is a less invasive alternative to endarterectomy to treat symptomatic or asymptomatic carotid stenosis. Large randomized clinical trials showed a higher periprocedural risk of non-disabling stroke with CAS and a higher periprocedural risk of myocardial infarction, cranial nerve palsy, and access site hematoma with CEA.

However little is known regarding the correlation between the morphological characteristics of the carotid plaque and the occurrence of microembolisation during the procedure and between microembolisation and midterm cognitive impairment. A few studies suggest that plaque morphology may be an important determinant for the increased risk of microembolisation. These studies however have mainly investigated microembolisation occurring during CAS and exploratory studies comparing the two procedures are still lacking.

The purpose of the present study is to determine the correlation between the morphological characteristics of the carotid plaque and cerebral microembolisation either after carotid stenting or after carotid endarterectomy in patients with symptomatic or asymptomatic carotid disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting a symptomatic (ipsilateral ischemic stroke, TIA located in the carotid artery territory or retinal ischemia) carotid stenosis between 50% and 99% (according to NASCET and ECST criteria)
* Patients presenting an asymptomatic carotid stenosis between 60% and 99% (according to NASCET and ECST criteria) Patients who accept the informed consent

Exclusion Criteria:

* Important neurological deficit with NIHSS >7 (or severe aphasia) at time of inclusion
* Previous known cognitive impairment
* Pregnancy
* Presence of contraindication based on ground of multidisciplinary team decision:

  * For surgery:

High bifurcation Intracranial extension of the carotid stenosis Patients with tandem lesions High suspicion of severe siphon stenosis Patients with previous irradiation of the cervical region Patients with restenosis after endarterectomy

* For stenting; Excessive arch vessel or carotid artery tortuosity and in particular presence tortuosity ≤90 degrees in the cervical segment Excessive aortic arch plaque burden Patients older than 70 years Unfavourable anatomic disposition as described above Co-morbidities that may preclude the use of a periprocedural dual antiplatelet regime.
* For CT-scan Iodine allergy Renal insufficiency
* For MRI Pacemaker Any other metallic implants Claustrophobia
* For ultrasound Bad quality ultrasound (patient morphology or equipments

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening of a carotid plaque is part of a routine procedure for patients admitted for stroke or TIA and includes ultrasound, CT-scan and MRI. Patients presenting a symptomatic or asymptomatic carotid stenosis are routinely discussed within a multidisciplinary meeting and the most appropriate therapeutic option is decided. For some patients, surgery and stenting are equivalent options. In that case, the patient may be a candidate for the present study
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Cerebral microembolisation | 24 hours
  the presence of at least 1 new hyperintense DWI lesion on the MRI realized within the 24 hours after procedure and will be correlated to the different characteristics of the carotid plaque evaluation.

SECONDARY OUTCOMES:
Neuropsychological assessment | 3 months
  Number and locations (watershed versus territorial) of the microembolisation will be dentified on DW-MRI and will be correlated to the neuropsychological changes after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Loraine Fisch, Principal Investigator — Junior consultant, neurovascular unit
Locations (1):
- Fisch Loraine, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murad MH, Coto-Yglesias F, Zumaeta-Garcia M, Elamin MB, Duggirala MK, Erwin PJ, Montori VM, Gloviczki P. A systematic review and meta-analysis of the treatments of varicose veins. J Vasc Surg. 2011 May;53(5 Suppl):49S-65S. doi: 10.1016/j.jvs.2011.02.031. PMID 21536173
- [Background] Bonati LH, Fraedrich G; Carotid Stenting Trialists' Collaboration. Age modifies the relative risk of stenting versus endarterectomy for symptomatic carotid stenosis--a pooled analysis of EVA-3S, SPACE and ICSS. Eur J Vasc Endovasc Surg. 2011 Feb;41(2):153-8. doi: 10.1016/j.ejvs.2011.01.001. Epub 2011 Jan 26. PMID 21269847
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Bonati LH, Jongen LM, Haller S, Flach HZ, Dobson J, Nederkoorn PJ, Macdonald S, Gaines PA, Waaijer A, Stierli P, Jager HR, Lyrer PA, Kappelle LJ, Wetzel SG, van der Lugt A, Mali WP, Brown MM, van der Worp HB, Engelter ST; ICSS-MRI study group. New ischaemic brain lesions on MRI after stenting or endarterectomy for symptomatic carotid stenosis: a substudy of the International Carotid Stenting Study (ICSS). Lancet Neurol. 2010 Apr;9(4):353-62. doi: 10.1016/S1474-4422(10)70057-0. Epub 2010 Feb 25. PMID 20189458
- [Background] Gensicke H, van der Worp HB, Nederkoorn PJ, Macdonald S, Gaines PA, van der Lugt A, Mali WP, Lyrer PA, Peters N, Featherstone RL, de Borst GJ, Engelter ST, Brown MM, Bonati LH; ICSS-MRI Substudy Investigators. Ischemic brain lesions after carotid artery stenting increase future cerebrovascular risk. J Am Coll Cardiol. 2015 Feb 17;65(6):521-9. doi: 10.1016/j.jacc.2014.11.038. PMID 25677309
- [Background] Rothwell PM, Slattery J, Warlow CP. Clinical and angiographic predictors of stroke and death from carotid endarterectomy: systematic review. BMJ. 1997 Dec 13;315(7122):1571-7. doi: 10.1136/bmj.315.7122.1571. PMID 9437274
- [Background] Biasi GM, Froio A, Diethrich EB, Deleo G, Galimberti S, Mingazzini P, Nicolaides AN, Griffin M, Raithel D, Reid DB, Valsecchi MG. Carotid plaque echolucency increases the risk of stroke in carotid stenting: the Imaging in Carotid Angioplasty and Risk of Stroke (ICAROS) study. Circulation. 2004 Aug 10;110(6):756-62. doi: 10.1161/01.CIR.0000138103.91187.E3. Epub 2004 Jul 26. PMID 15277320
- [Background] Varetto G, Gibello L, Faletti R, Gattuso A, Garneri P, Castagno C, Quaglino S, Rispoli P. Contrast-enhanced ultrasound to predict the risk of microembolization during carotid artery stenting. Radiol Med. 2015 Nov;120(11):1050-5. doi: 10.1007/s11547-015-0530-4. Epub 2015 Mar 25. PMID 25805183
- [Background] Maggio P, Altamura C, Landi D, Migliore S, Lupoi D, Moffa F, Quintiliani L, Vollaro S, Palazzo P, Altavilla R, Pasqualetti P, Errante Y, Quattrocchi CC, Tibuzzi F, Passarelli F, Arpesani R, di Giambattista G, Grasso FR, Luppi G, Vernieri F. Diffusion-weighted lesions after carotid artery stenting are associated with cognitive impairment. J Neurol Sci. 2013 May 15;328(1-2):58-63. doi: 10.1016/j.jns.2013.02.019. Epub 2013 Mar 17. PMID 23510565
- [Background] Yun TJ, Sohn CH, Han MH, Yoon BW, Kang HS, Kim JE, Paeng JC, Choi SH, Kim JH, Chang KH. Effect of carotid artery stenting on cerebral blood flow: evaluation of hemodynamic changes using arterial spin labeling. Neuroradiology. 2013 Feb;55(3):271-81. doi: 10.1007/s00234-012-1104-y. Epub 2012 Oct 24. PMID 23093072